CLINICAL TRIAL: NCT03633708
Title: Phase 3, Randomized, Open-label, Controlled, Multiple Dose, Efficacy, Safety, Pharmacokinetic, and Pharmacodynamic Study of Etelcalcetide in Pediatric Subjects 28 Days to < 18 Years of Age With Secondary Hyperparathyroidism and Chronic Kidney Disease Receiving Maintenance Hemodialysis
Brief Title: A Study of Etelcalcetide in Pediatric Subjects With Secondary Hyperparathyroidism and Chronic Kidney Disease on Hemodialysis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140315; 2017-002411-34 (EudraCT Number)
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease
Keywords: sHPT; CKD; pediatric; Secondary Hyperparathyroidism; Chronic Kidney disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etelcalcetide (Experimental): Randomized in a 3:1 ratio to receive etelcalcetide in addition to standard of care
  Interventions: Drug: Etelcalcetide
- Control (Active Comparator): Randomized in a 3:1 ratio to receive etelcalcetide in addition standard of care alone (control arm)
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Etelcalcetide has been shown to be safe and efficacious in treating adult CKD patients with SHPT by simultaneously controlling intact parathyroid hormone (iPTH), Ca, and phosphorus and has recently been approved for use in adult patients with SHPT treated with hemodialysis in both the United States and Europe
  Other Names: Parsabiv

SUMMARY:
This is a Phase 3 Study of Etelcalcetide in Pediatric Subjects With Secondary Hyperparathyroidism and Chronic Kidney Disease on Hemodialysis

DETAILED DESCRIPTION:
SHPT is a common and serious co-morbidity that develops relatively early in the course of CKD, worsens with declining kidney function, and is associated with serious complications in children on dialysis. Children on dialysis experience a wide spectrum of bone abnormalities and growth retardation, in addition to increased risk for cardiovascular morbidity and mortality that manifests early in their adulthood. Traditional therapies for SHPT (eg, vitamin D sterols) are widely used in the pediatric dialysis population, and have the potential to aggravate complications of the disease by increasing serum calcium (Ca), serum phosphorus, and serum Ca times serum phosphorus product.

Etelcalcetide has been shown to be safe and efficacious in treating adult CKD patients with SHPT by simultaneously controlling intact parathyroid hormone (iPTH), Ca, and phosphorus and has recently been approved for use in adult patients with SHPT treated with hemodialysis in both the United States and Europe. Although no previous studies have been conducted in pediatric patients with etelcalcetide (one single dose pharmacokinetic [PK] study is currently ongoing),Amgen anticipates minimal to moderate risk with a possibility of direct benefit to the pediatric subjects (age 28 days to 18 years) in this study. The burden of complications of SHPT in the pediatric dialysis population and the limitations of current standard therapy, underscore the need for studies of etelcalcetide in these patients to address this unmet medical need and inform the pediatric nephrology community of the potential use of etelcalcetide in children on hemodialysis with critical safety and efficacy data.

ELIGIBILITY:
Inclusion criteria

* Age of 28 days or older and less than 18 years
* Dry weight ≥ 7 kg during screening.
* Diagnosed with CKD and SHPT undergoing hemodialysis at the time of screening.
* Diagnosis of SHPT with the mean of the 2 consecutive central laboratory iPTH values ≥ 400 pg/mL (42 pmol/L) during screening, on separate days and within 2 weeks of enrolment.
* Serum cCa value ≥ 9.0 mg/dL (2.25 mmol/L) for subjects ≥ 2 years of age and older and serum cCa value ≥ 9.6 mg/dL (2.4 mmol/L) for subjects 28 days to < 2 years of age obtained from the central laboratory during screening.
* Dialysate Ca level ≥ 2.5 mEq/L during screening for at least 4 weeks prior to screening and throughout the duration of the study.
* No more than a maximum prescribed dose change of 50% for active vitamin D sterols/phosphate binders/Ca supplements within the 2 weeks prior to screening assessments and remain stable.
* SHPT not due to vitamin D deficiency, per investigator assessment.

Exclusion Criteria Disease Related

* History of congenital long QT syndrome, second or third degree heart block, ventricular tachyarrhythmia's or other conditions associated with prolonged QT interval.
* Anticipated or scheduled parathyroidectomy during the study period.
* Anticipated or scheduled kidney transplant during the study period.
* Subject has received a parathyroidectomy within 6 months prior to randomization.

Other Medical Conditions

* History of other malignancy, except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within the last 5 years. Prior/Concomitant Therapy
* Use of concomitant medications that may prolong the corrected QT interval (eg, ondansetron, albuterol, sotalol, amiodarone, erythromycin, or clarithromycin). Refer to CredibleMeds.org for guidance.
* Receipt of cinacalcet therapy within 30 days prior to screening assessments and through randomization.
* Receipt of etelcalcetide within 6 months prior to screening assessments and through randomization.
* All herbal medicines (eg, St. John's wort), vitamins, and supplements consumed by the subject within the 30 days prior to randomization, and continuing use if applicable, will be reviewed by the Principal Investigator and the Amgen Medical Monitor. Written documentation of the review and Amgen acknowledgment is required for subject participation.
* Use of any over-the-counter or prescription medications within the 14 days or 5 half-lives (whichever is longer) prior to randomization that are not established therapies for subjects with renal disease or other conditions secondary to renal disease will be reviewed by the Principal Investigator and the Amgen Medical Monitor. Written documentation of the review and Amgen acknowledgment is required for subject participation. Paracetamol for analgesia will be allowed.

Prior/Concurrent Clinical Study Experience • Currently receiving treatment in another investigational device or drug study, or less than 30 days or 5 half-lives (whichever is longer) since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.

Diagnostic Assessments During Screening

* Subject has significant abnormalities on the most recent central laboratory test during the screening period prior to enrollment per the Investigator including but not limited to the following: a. Serum transaminase (alanine aminotransferase [ALT] or serum glutamic pyruvic transaminase [SGPT], aspartate aminotransferase [AST] or serum glutamic oxaloacetic transaminase [SGOT]) > 2.0 times the upper limit of normal (ULN).
* Corrected QT interval (QTc) > 500 ms, using Bazett's formula.
* QTc ≥ 450 to ≤ 500 ms, using Bazett's formula, unless written permission to enroll is provided by the investigator after consultation with a pediatric cardiologist.
* Subject has a clinically significant electrocardiogram (ECG) abnormality during screening that, in the opinion of the investigator, could pose a risk to subject safety or interfere with the study evaluation.

Within the 60 days prior to enrollment

• New onset or worsening of a pre-existing seizure disorder.

Other Exclusions

* Subjects aged 28 days to 6 months of age who were born prematurely at < 36 weeks gestational age.
* Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 3 months after the last dose of etelcalcetide. (Females of childbearing potential should only be included in the study after a confirmed menstrual period and a negative highly sensitive serum pregnancy test within 7 days prior to the first dose of investigational product).
* Female subjects of childbearing potential unwilling to use 1 highly-effective or acceptable method of contraception during treatment and for an additional 3 months after the last dose of investigational product.
* Subject has known sensitivity to etelcalcetide or excipients to be administered during dosing.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, to the best of the subject and investigator's knowledge).
* History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Subject has previously entered this study

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with ≥ 30% reduction from baseline in intact parathyroid hormone (iPTH) level during the efficacy assessment phase (EAP) | Baseline and Weeks 20-27
  Achievement of at least a 30% reduction from baseline in mean iPTH during the EAP (defined as weeks 20 through 27).

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of etelcalcetide | 10-30 minutes post dose on Day 1 and 10-30 minutes post dose on Weeks 5, 9, 13, 17, and 21
  Cmax will be collected and reported for the etelcalcetide arm only.
Minimum serum concentration (Cmin) of etelcalcetide | 10-30 minutes post dose on Day 1 and 10-30 minutes post dose on Weeks 5, 9, 13, 17, and 21
  Cmin will be collected and reported for the etelcalcetide arm only.
Incidence of adverse events | Day 1 to 30 days after last dose of etelcalcetide (up to approximately 30 weeks)
  To characterize the safety of etelcalcetide treatment based on adverse events. Nature, frequency, severity, and relationship to treatment of all adverse events, including those of special interest reported during the study.
Frequency of hypocalcemia | Up to approximately 30 Weeks
  Occurrence of hypocalcemia at any point in time, assessed by serum chemistry.
Number of participants with corrected serum calcium levels at any time during the study | Up to approximately 30 Weeks
  Occurrence of corrected serum Ca levels <8.0 mg/dL (2.0 mmol/L) for subjects 2 to < 18 years of age and <8.6 mg/dL (2.15 mmol/L) for subjects 28 days to <2 years of age during the study.
Number of participants with serum phosphorous levels below normal for age | Up to approximately 30 Weeks
  Occurrence of serum phosphorous levels below the lower limit of normal for age.
Number of participants with predialysis iPTH levels below normal | Up to approximately 30 Weeks
  Occurrence of predialysis iPTH levels below the lower limit of normal for age.
Change from baseline in systolic blood pressure | Week -2, Week -1, Day1, and Weeks 4, 8, 12, 16, 20, 24, and 27
  To characterize the safety of etelcalcetide treatment based on vital signs.
Change from baseline in diastolic blood pressure | Week -2, Week -1, Day1, and Weeks 4, 8, 12, 16, 20, 24, and 27
  To characterize the safety of etelcalcetide treatment based on vital signs.
Change from baseline in heart rate | Week -2, Week -1, Day1, and Weeks 4, 8, 12, 16, 20, 24, and 27
  To characterize the safety of etelcalcetide treatment based on vital signs.
Change in Tanner Stage | Week -2 and Week 27
  Changes in tanner stage at scheduled visits.
Change in height | Day 1 and Week 27
  Changes in height at scheduled visits.
Change in weight | Week -2, Day 1, and Week 27
  Changes in weight at scheduled visits.
Achievement of ≥ 30% reduction in iPTH from baseline on two consecutive visits | Up to approximately 30 Weeks
  To characterize change in laboratory markers of CKD following etelcalcetide treatment.
Mean change from baseline in predialysis iPTH | Baseline and Weeks 20-27
  Mean change from baseline in predialysis iPTH during the EAP (defined as weeks 20 through 27).
Percentage change from baseline in predialysis iPTH | Baseline and Weeks 20-27
  Percentage change from baseline in predialysis iPTH during the EAP (defined as weeks 20 through 27).
Percentage change from baseline in corrected total serum calcium | Baseline and Weeks 20-27
  Percentage change from baseline in corrected total serum calcium during the EAP (defined as weeks 20 through 27).
Percentage change from baseline in corrected total serum phosphorous | Baseline and Weeks 20-27
  Percentage change from baseline in corrected total serum phosphorous during the EAP (defined as weeks 20 through 27).

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (43):
- United States (10):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Childrens Mercy Hospital, Kansas City, Missouri
  - Mount Sinai Kidney Center - B1 Renal Treatment, New York, New York
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Childrens Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Medical Center Dallas, Dallas, Texas
  - Primary Childrens Hospital Outpatient Services, Salt Lake City, Utah
- Argentina (3):
  - Fresenius Escobar, Belén de Escobar, Buenos Aires
  - Hospital Italiano, Cuidad Autonoma de Buenos Aires, Buenos Aires
  - Centro Infantil Del Rinon, San Miguel de Tucumán, Tucumán Province
- India (6):
  - Manipal Hospital, Bangalore, Karnataka
  - KLES Dr Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - Fortis Flt Lt Rajan Dhall Hospital, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - NRS Medical College and Hospital, Kolkata, West Bengal
- Malaysia (3):
  - Hospital Raja Perempuan Zainab II, Kota Bharu, Kelantan
  - Hospital Wanita Dan Kanak-Kanak Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - Hospital TuanKu Jaafar, Seremban, Negeri Sembilan
- Russia (3):
  - SBHI Pediatrics city clinical hospital of Saint Vladimir, Moscow
  - SBHI Children's City Multidisciplinary Clinical Specialized Center of High Medical Technologies, Saint Petersburg
  - State Budgetary Healthcare Institution Samara Regional Clinical Hospital na V D Seredavin, Samara
- National University Hospital, Singapore, Singapore
- South Korea (3):
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Pusan National University Yangsan Hospital, Yangsan-si, Gyeongsangnam-do
- Taiwan (4):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (9):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Baskent Universitesi Ankara Hastanesi, Ankara
  - Gazi Universitesi Saglik Arastirma ve Uygulama Merkezi Gazi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Firat Universitesi Tip Fakultesi Hastanesi, Elâzığ
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Marmara Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Erciyes Universitesi Tip Fakultesi Hastanesi, Kayseri
- National Childrens Specializated Hospital Okhmadit, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com